CLINICAL TRIAL: NCT01340248
Title: A Randomized, Open-label, Single-dose, Crossover Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics of Dilatrend SR 64mg Capsule After Oral Administration in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Chong Kun Dang Pharmaceutical, Cho, Jung Ah/CRA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 125HPS11F
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Stable Angina
Keywords: food effect; pharmacokinetics; healthy male volunteers
MeSH Terms: conditions — Angina, Stable | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dilatrend 64mg capsule (Experimental): * Randomized, open-label, single dose, two-period, two-way, crossover study
  1. group : Dilatrend 64mg capsule during fasting + Dilatrend 64mg capsule after high fat diet
  2. group : Dilatrend 64mg capsule after high fat diet + Dilatrend 64mg capsule during fasting
  Interventions: Drug: Dilatrend 64mg capsule

INTERVENTIONS:
Drug: Dilatrend 64mg capsule — 1. Dilatrend 64mg capsule during fasting + Dilatrend 64mg capsule after high fat diet
  2. Dilatrend 64mg capsule after high fat diet + Dilatrend 64mg capsule during fasting

SUMMARY:
A randomized, open-label, single-dose, crossover clinical trial to evaluate the food effect on the pharmacokinetics of Dilatrend SR 64mg capsule after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 50 aged in healthy adults
* Weight more than 55kg, IBW 20% within the range
* Agreement with written informed consent

Exclusion Criteria:

* Subject has hypersensitivity reaction or clinically significant history about investigational drug
* Clinically significant cardiovascular system, respiratory system, liver, renal, endocrine system, gastrointestinal system, central nervous system, blood tumor, mental disease, skin disease and so on
* Inadequate result of laboratory test

  * AST(SGOT) or ALT(SGPT) > 1.5 x upper limit of normal range
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 210 g/day) or during clinical trials can not be drunk or severe heavy smoker (cigarette > 10 cigarettes per day)
* Creatinine clearance < 80ml/min
* Subject with known for history(such as gastrointestinal disease or operation) with affect the absorption of drug
* Subject takes an abnormal meal which affect the ADME of drug
* Previously participated in other trial within 90 days
* Previously make whole blood donation within 60 days or component blood donation within 30 days
* Subject with positive reaction for reason of laboratory test result
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
evaluation of pharmacokinetics | pre-dose(0h), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48h
  The effect of food on PK after high fat diet and fasting Blood sampling over a 72 hour period post dose in all dosing sessions

SECONDARY OUTCOMES:
evaluation of safety | from screenig to post-study visit
  * adverse event monitoring
  * physical examination, vital sign, ECOG, laboratory test

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university, Daegu, Seoul, South Korea